CLINICAL TRIAL: NCT00394797
Title: Surgical Correction of Moderate Ischemic Mitral Regurgitation
Status: Completed | Type: Observational
Sponsor: Shaare Zedek Medical Center (Other)
Other Study IDs: IMR001
Record Dates: First submitted 2006-10-31; First posted 2006-11-01 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2011-05

CONDITIONS: Moderate Ischemic Mitral Regurgitation
MeSH Terms: interventions — Mitral Valve Annuloplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Procedure: mitral valve annuloplasty

SUMMARY:
The purpose of this study is to try and determine whether repair of moderate ischemic mitral regurgitation at the time of coronary bypass graft surgery (CABG) has an impact on survival.We will compare patients undergoing CABG + mitral repair or CABG only groups. Primary endpoints include late survival. Secondary endpoints include event free survival, symptoms, and echocardiographic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing coronary bypass surgery who have moderate degree of ischemic MR

Exclusion Criteria:

* etiology of mitral regurgitation other than ischemic, degree of regurgitation other than moderate.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing coronary bypass surgery who have moderate degree of ischemic MR
Sampling Method: Probability Sample

PRIMARY OUTCOMES:
survival at 1,5 and 10 years

SECONDARY OUTCOMES:
event free survival
symptoms
echocardiographic parameters

CONTACTS AND LOCATIONS:
Overall Officials: Shuli Silberman, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel